CLINICAL TRIAL: NCT03964909
Title: Resting-State Functional MRI in Glioma Patients Before and After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0906; NCI-2019-02653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0906 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Brain Mass; Glioma
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (fMRI, CVR MRI, rs-fMRI) (Experimental): Patients undergo standard of care fMRI, CVR MRI over 3 minutes, and rs-fMRI over 6 minutes 1 month before and within 6 weeks after standard of care surgery.
  Interventions: Procedure: Functional Magnetic Resonance Imaging; Procedure: Magnetic Resonance Imaging; Procedure: Resting State Functional Connectivity Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Functional Magnetic Resonance Imaging — Undergo fMRI
  Other Names: fMRI; Functional MRI
Procedure: Magnetic Resonance Imaging — Undergo CVR MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Resting State Functional Connectivity Magnetic Resonance Imaging — Undergo rs-fMRI
  Other Names: Resting fcMRI; Resting State Functional Connectivity MRI; RS-fcMRI

SUMMARY:
This clinical trial studies how well resting-state functional magnetic resonance imaging (MRI) and cerebrovascular reactivity (CVR) MRI performed before and after surgery works in measuring the effects on language in patients with glioma. Mapping language function before brain tumor resection is crucial for preventing post-surgical deficits and maximizing restoration of language function following surgery. Additional imaging, such as resting-state functional MRI and CVR MRI, may help measure the language network in the brain before surgery and any effects on language function after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a reliable platform for preoperative mapping of language networks using resting-state-functional magnetic resonance imaging (rs)-fMRI in glioma patients.

SECONDARY OBJECTIVES:

I. To explore the reorganizations of resting-state functional connectivity (FC) and their relation to neuropsychological outcomes in glioma patients after surgery.

OUTLINE:

Patients undergo standard of care functional (f)MRI, CVR MRI over 3 minutes, and rs-fMRI over 6 minutes 1 month before and within 6 weeks after standard of care surgery.

After completion of study, patients are followed up at 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed brain mass suspected to be gliomas
* English speaker
* Right handed
* Tumor is located on or adjacent to Broca's or Wernicke's areas in the hemisphere suspected to be dominant for language
* No prior history of neurologic disease or insult, or neuropsychiatric illness requiring treatment that would affect cognition in the opinion of the attending neuropsychologist
* Patients who will undergo neurosurgical resection
* Patients who are on neurosurgical evaluation will undergo direct cortical stimulation (DCS) as standard of care
* Patients who will complete pre- and postoperative neuropsychological testing per standard of care
* Pregnant women

Exclusion Criteria:

* Patients with prior radiation or chemotherapy
* Patients cannot give informed consent
* Patients cannot undergo MRI and functional MRI examinations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Detectability of language networks | Up to 6 weeks
  Will be performed using resting-state-functional magnetic resonance imaging (rs-fMRI). The receiver operating characteristic (ROC) analysis will be carried out to compare the difference between the diagnostic performance of the proposed method and that of the data-driven rs-fMRI method. The study will evaluate the performance of rs-fMRI by comparing with the standard of care intraoperative direct cortical stimulation.

SECONDARY OUTCOMES:
Changes in resting-state functional connectivity and neuropsychological outcomes | Up to 6 weeks
  Graph theoretical analysis and large-scale network analysis will be applied to analyze pre- and post- surgical rs-fMRI data, to explore how the functional reorganization is correlated to the changes of neuropsychological scores. Correlational analyses will be conducted to determine the associations between changes in rs-fMRI network features and neuropsychological functioning from the pre- to postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Ling A Liu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org